CLINICAL TRIAL: NCT04372732
Title: Clinical Study on the Role of New Serum Tumor Autoantibodies in Predicting the Efficacy of Anti-PD-1 Immunotherapy in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Serum Autoantibodies in Predicting the Efficacy of Anti-PD-1 Treatment in Patients With Advanced NSCLC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chang Chen, PhD,MD, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: K20-188
Record Dates: First submitted 2020-04-27; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer; Immunotherapy
Keywords: PD-1/PD-L1 blockades; tumor autoantiboby; NSCLC; predictive factor; prognosis; immunotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: All participants will be detected for antoantibodies and then treated with PD-1 blockade.
  Interventions: Diagnostic Test: Serum tumor autoantibody detection

INTERVENTIONS:
Diagnostic Test: Serum tumor autoantibody detection — All enrolled patients will be tested for ten kinds of tumor autoantibodies using peripheral blood before PD-1 bloackade treatment.

SUMMARY:
PD-1/PD-L1 blockades have attracted much attention in the treatment of lung cancer, however only a small set of patients can benefit from this kind of immunotherapy. At present, the expression level of PD-L1 is the major factor to evaluate the prognosis，, which is highly dependent on the quality of tissue samples and detection methods.Therefore, finding predictive markers,especially based on liquid biopsy, to screen the patients who will benefit most from PD-1/PD-L1 blockades is an urgent issue in immunotherapy for lung cancer. Tumor autoantibodies, as immune response products of the immune system to tumor antigens, are of great significance in tumor diagnosis. Till now, the relationship between tumor autoantibodies and immunotherapy efficacy has not been reported. In this study, 200 non-small cell lung cancer patients will be enrolled with baseline serum tumor autoantibodies detection, then treated with PD-1 blockade. The purpose of this study is to explore the correlations of serum autoantibodies expression and efficacy of PD-1 inhibitor, so that to identify new markers for predicting the efficacy of PD-1/PD-L1 immunotherapy in non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects understood the requirements and risks of the study fully and signed the informed consent form.
2. Aged between 18 and 70 years;
3. Histologically or cytologically confirmed diagnosis of advanced non-small cell lung cancer.
4. Immunohistochemistry of pathological tissue: PD-L1 (22C3) ≥ 1%,Gene detection EGFR (-); ALK (-), ROS1 (-).
5. All of these patients have no surgical indications or radical radiotherapy guidelines.
6. ECOG PS score 0-1, life expectancy not less than 12 weeks.
7. According to RECIST1.1,there is at least one tumor site that can be accurately measured by CT in patients.
8. Women of childbearing age had negative pregnancy tests and were willing to accept drugs or intrauterine contraception, while men of childbearing age were willing to accept contraception voluntarily.
9. Adequate hematologic function:Peripheral blood neutrophil count > 2000 cells / uL, Platelet count > 100*109 / L; Hemoglobin >9.0g/dL;Blood total bilirubin < 2 times normal upper limit, blood AST and ALT ≤ 2. 5 times normal upper line;Inosine clearance ≥ 60ml / min.

Exclusion Criteria:

1. Subjects who needed to receive systemic corticosteroids (prednisone equal to or higher than 10mg / day) or other immunosuppressive drugs within 14 days before enrollment or during the study.
2. Subjects who had been vaccinated with antineoplastic vaccine or received antineoplastic drugs with immunostimulatory effect within 4 weeks before entering the group.
3. Subjects with known or suspected active autoimmune diseases (vitiligo, type I diabetes, autoimmune thyroiditis requiring hormone replacement therapy, and other autoimmune diseases without recurrence can also be included).
4. Subjects with other tumors in the past 5 years, except cervical carcinoma in situ, basal cell carcinoma of the skin, etc.
5. Subjects with any unstable systemic diseases (including active infections, poorly controlled hypertension, unstable angina pectoris, angina pectoris that occurred in the past 3 months, congestive heart failure (or New York Heart Association (NYHA) II)), infarcts (within 6 months), severe arrhythmias requiring medication, liver, kidney or metabolic diseases.
6. Subjects with previous or present interstitial lung diseases.
7. Subjects with systemic infection who need to be treated, HBV surface antigen positive or HCV RNA positive; patients who have previously or currently detected human immunodeficiency virus (HIV) or AIDS.
8. Subjects who received targeted therapy or biotherapy at the same time.
9. Subjects who are allergic to therapeutic drugs (chemotherapeutic drugs and immune drugs);
10. Subjects who underwent major surgery or suffered severe trauma within 2 months before the first treatment;
11. Situations that other researchers do not consider appropriate to be included.
12. Subjects whose expected survival time is less than 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced non-small cell lung cancer, PD-L1 expression ≥1%, EGFR/ALK/ROS1 wild type will be studied. The serum autoantibodies will be detected before PD-1 blockade treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
The correlations of tumor autoantibodies and PFS/ORR of PD-1 blockade treatment. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To analyze the relationships of serum tumor autoantibody expression and PFS (progression-free survival) and ORR ( objective response rate) of enrolled patients treated with PD-1 blockade.

SECONDARY OUTCOMES:
The correlations of tumor autoantibodies and OS/DCR of PD-1 blockade treatment. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To analyze the relationships of serum tumor autoantibody expression and OS (overall survival) and DCR (disease control rate) of enrolled patients treated with PD-1 blockade.